CLINICAL TRIAL: NCT00165243
Title: Tangential Radiation Therapy Without Axillary Dissection in Early-Stage Breast Cancer
Brief Title: Tangential Radiation Therapy Without Axillary Dissection in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Julia S. Wong, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98-101
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Early-Stage Breast Cancer
Keywords: Axillary Dissection; Tangential Radiation; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Tangential radiation — Radiation given over 6 1/2 weeks

SUMMARY:
The purpose of this study is to evaluate whether treatment to the axilla (area under the arm) can be safely minimized by omitting axillary surgery and full axillary radiation therapy and replacing it with radiation therapy to the breast and lower axilla.

DETAILED DESCRIPTION:
* Patients will have undergone conservative breast surgery without axillary dissection prior to enrollment in this study.
* Patients will receive radiation therapy to the breast, including the lowest axillary lymph nodes, over a period of 6 1/2 weeks.
* No radiation will be specifically directed toward the upper axilla or supraclavicular lymph nodes.
* Patients will also receive 5 years of tamoxifen or another type of hormone therapy determined by the medical oncologist.
* Follow-up visits will occur every 6 months and mammograms every 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinical stage I or II breast cancer, clinically uninvolved axillary nodes.
* Patients must be 55 years or older.
* Patients must undergo total excision of the primary invasive tumor
* Final pathologic margin status must be negative
* Only estrogen receptor (ER) or progesterone receptor (PR) positive tumors will be permitted

Exclusion Criteria:

* Prior history of malignancy, except for non-melanoma skin cancers and carcinoma in situ fo the cervix

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1998-09; Primary Completion 2004-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To determine if patients with early-stage breast tumors can be effectively treated by tangential breast radiation. | 5 years

SECONDARY OUTCOMES:
To determine the safety of this treatment. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Julia S. Wong, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts